CLINICAL TRIAL: NCT06341205
Title: Study of Artificial Intelligence-based Personalized Rituximab Treatment Protocol in Membranous Nephropathy
Brief Title: Personalized Rituximab Treatment Based on Artificial Intelligence in Membranous Nephropathy (iRITUX)
Acronym: iRITUX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-APN-01
Record Dates: First submitted 2024-02-27; First posted 2024-04-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard-of-care (Active Comparator): rituximab treatment 1gram x 2 (day-0, day-15)
  Interventions: Drug: RiTUXimab Injection
- Personalised treatment (Experimental): personalized treatment based on the algorithm for assessing the risk of having undetectable rituximab level after 3 months:
  * Patients with a risk between 0 and 50% will receive 1gram x2 (day-0, day-15)
  * Patients with a risk between 51 and 75% will receive 1gram x 3 (day-0, day-15, day-30)
  * Patients with a risk between 76 and 100% will receive 1gram x 4 (day-0, day-15, day-30, day-45)
  Interventions: Drug: RiTUXimab Injection

INTERVENTIONS:
Drug: RiTUXimab Injection — Dose administered will depend on randomisation and for experimental Arm on the risk of having undetectable rituximab level after 3 months

SUMMARY:
Membranous nephropathy is an autoimmune disease affecting the kidney, and the most common cause of nephrotic syndrome in non-diabetic Caucasian adults. The course of this disease is highly variable from one individual to another, ranging from spontaneous remission to progressive chronic kidney disease.

The identification of autoantibodies - e.g., the phospholipase A2 receptor type 1 (PLA2R1) - has promoted the use of immunosuppressive drugs such as rituximab which is now a safe and effective first-line treatment for the management of membranous nephropathy. However, up to 40% of patients do not respond to a first course of rituximab treatment. In nephrotic patients, due to urinary drug loss, rituximab blood level is lower than in other autoimmune diseases treated with rituximab without proteinuria. This high urinary drug loss decreases the drug exposure, potentially explaining why rituximab regimen with low dose infusions (375 mg/m2) did not demonstrate efficacy after month-6 compared to a non-immunosuppressive antiproteinuric treatment in a previous study. In contrast, a regimen of two 1-g infusions two weeks apart was associated with a significantly greater remission rate after 6 months.

Recently, the investigators have shown that after two 1-g rituximab infusions, the rituximab blood level 3 months after the first rituximab infusion, was correlated with the likelihood of remission after 6 and 12 months of the rituximab treatment. Patients with positive rituximab blood level 3 months after treatment had a higher chance of remission at month-6 and at month-12 than patients with an undetectable rituximab level at month-3.

Nowadays, machine learning algorithms are increasingly used in medicine, especially in pharmacology, to predict the exposure to a drug, the initial dose to administer or the interval between two infusions.

The objective of this study is to use a machine learning algorithm predicting the risk of having an undetectable residual level of rituximab 3 months after treatment, in order to propose a personalized treatment management with early additional doses of rituximab for the patients at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ongoing episode of membranous nephropathy diagnosed by the presence of anti-PLA2R1 antibodies detected by ELISA (≥ 14 RU/ml, EUROIMMUN): the result must be validated by the Coordination team before randomization.
* Nephrotic syndrome defined by proteinuria > 3.5 g/24h (or UPCR > 3.5 g/g) and serum albumin < 30 g/L at diagnosis
* Estimated Glomerular Filtration Rate (CKD-EPI formula) > 30 mL/min/1,73 m2
* Indication for rituximab treatment according to the KDIGO and French guidelines
* Non-immunosuppressive antiproteinuric treatment at stable dose for 2 weeks according to French guidelines, including a renin angiotensin aldosterone system inhibitor, a diuretic and a low-salt diet at maximal tolerated dose (i.e., absence of orthostatic hypotension and no increase in creatinine > 30%)

Exclusion Criteria:

* Secondary Membranous nephropathy related to cancer, infection, systemic lupus, drug
* Diagnosis of PLA2R1-associated Membranous nephropathy not confirmed by the Coordination team (validation mandatory for randomization)
* Pregnancy or breastfeeding
* Immunosuppressive treatment (including rituximab) in the 6 months preceding inclusion
* Presence of anti-rituximab antibodies detected by Central Lab
* Cancer under treatment
* Patients with active, severe infections
* Hypersensitivity to the active substance or excipients
* Patients severely immunocompromised
* Severe heart failure or severe, uncontrolled cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2031-08-31 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission (complete or partial) after 6 months of rituximab initiation | 6 months
  Clinical remission (complete or partial) according to KDIGO and French guidelines:
  * Complete: urine protein/creatinine ratio (UPCR) <0.3 g/g and serum albumin>30 g/L and Glomerular Filtration Rate (estimated by CKD-EPI formula) >60 ml/min/1.73m2
  * Partial: UPCR <3.5 g/g with a decrease >50% from baseline (i.e., at first rituximab infusion) and serum albumin improvement or normalization and stable serum creatinine (or increase <30%).

SECONDARY OUTCOMES:
Complete clinical remission after 12 months of rituximab initiation | 12 months
  Complete remission: urine protein/creatinine ratio (UPCR) <0.3 g/g and serum albumin>30 g/L and Glomerular Filtration Rate (estimated by CKD-EPI formula) >60 ml/min/1.73m2
Partial clinical remission after 12 months of rituximab initiation | 12 months
  Partial remission: UPCR <3.5 g/g with a decrease >50% from baseline (i.e., at first rituximab infusion) and serum albumin improvement or normalization and stable serum creatinine (or increase <30%).
Immunological remission: anti-PLA2R1 depletion | 12 months
  Immunological remission: anti-PLA2R1 depletion (i.e., PLA2R1 titer < 14 RU/mL by ELISA method) at month-3, month-6 and month-12
Change in urine protein/creatinine ratio (UPCR) | 12 months
  Percentage of change in urine albumin/creatinine ratio (mg/g) from day-0 to month-3, month-6, month-9, month-12
Change in serum creatinine | 12 months
  Percentage of change in serum creatinine (μmol/L) from day-0 to month-3, month-6, month-9, month-12
Change in renal function | 12 months
  Percentage of change in Glomerular Filtration Rate estimated by CKD-EPI formula (mL/min/1.73m²) from day-0 to month-3, month-6, month-9, month-12
Change in the immunological status of the disease | 12 months
  Percentage of change in anti-PLA2R1 titer (RU/mL) by ELISA (EUROIMMUN Kit) from day-0 to month-3, month-6, month-9, month-12
Appearance of anti-drug antibodies after rituximab treatment | 12 months
  Serum anti-rituximab antibodies (ng/mL) at month-3, month-6, month-9, month-12
Rituximab underdosed patients | 3 months
  Percentage of patients with serum rituximab (μg/mL) >2 μg/mL 3 months after the last infusion
Serious adverse events | 84 months
  Occurence of Serious adverse events reported
Adaptation of symptomatic treatment | 84 months
  Number of dose modification of non-immunosuppressive anti-proteinuric treatment during study follow-up
Model improvement through machine learning | 6 months
  serum creatinine and serum albumin levels, weight, anti-PLA2R1 and rituximab level will be combined to report the risk of having undetectable rituximab level after 3 months (in %) at day-0, day-15, day-30, day-45, month-3, month-6
Effect of rituximab on immune profiles | 6 months
  Cytokine levels in pg/mL (IFN-γ, IFN-α, IL-12p70, IL-17A, IL-4, IL-5, IL-10, IL-1, IL-6) at day-0 and month-6

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU de BESANCON, Besançon
  - CHU de BORDEAUX - Hôpital Pellegrin, Bordeaux
  - CHU de CAEN, Caen
  - AP-HP - Hôpital H. Mondor, Créteil
  - HCL - Hôpital E. Herriot, Lyon
  - AP-HM - Hôpital de la Conception, Marseille
  - CHU de NICE, Nice
  - CHU de Nîmes - Hôpital CAREMEAU, Nîmes
  - AP-HP - Hôpital Européen Georges Pompidou, Paris
  - AP-HP - Hôpital Necker, Paris
  - CHU de TOULOUSE - Hôpital Rangueil, Toulouse
  - CHRU de TOURS - Hôpital Bretonneau, Tours
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No
not planed

REFERENCES:
- [Derived] Teisseyre M, Destere A, Cremoni M, Zorzi K, Brglez V, Benito S, Bailly L, Fernandez C, Seitz-Polski B. Artificial intelligence-based personalised rituximab treatment protocol in membranous nephropathy (iRITUX): protocol for a multicentre randomised control trial. BMJ Open. 2025 Apr 2;15(4):e093920. doi: 10.1136/bmjopen-2024-093920. PMID 40180405